CLINICAL TRIAL: NCT05740826
Title: Correlation Between Cervical Spine Muscle Disorders and the Occurrence of Symptoms of Temporomandibular Joint Dysfunction
Status: Completed | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jagoda Goślińska, Dr Jagoda Goślińska, Poznan University of Medical Sciences
Other Study IDs: 676/22
Record Dates: First submitted 2023-02-10; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Temporomandibular Joint Disorders
Keywords: TMJ disorders; pressure sensitivity; algometer; young adults; myofascial pain
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: People with temporomandibular disorder which was determined based on one of the following factors observed during the examination: acoustic symptoms, present temporomandibular joint pain, problems with opening the mouth, deviation of the jaw during abduction, or reported locking of the jaw.
  Interventions: Device: Algometer
- Control group: People without temporomandibular disorder.
  Interventions: Device: Algometer

INTERVENTIONS:
Device: Algometer — The algometer head was applied to the trigger point of selected muscles at an angle of 90° and, increasing the pressure at a speed of about 100g/s, three measurements were made. Each measurement stoped at the first sensation of pain

SUMMARY:
This study evaluated the correlation between the occurrence of disorders of selected muscles of the cervical spine and the occurrence of symptoms of TMJ dysfunction

DETAILED DESCRIPTION:
The examination includes personal questionnaire, physical examination and an algometer measurement on the upper fibers of the trapezius, levator scapula, sternocleidomastoid and rectus capitis posterior major to define pressure sensitivity of neck muscles and define is there a correlation between the occurrence of disorders of selected muscles of the cervical spine and the occurrence of symptoms of TMJ dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* age 19-25 years
* relatively good health
* consent to participate in the research experiment

Exclusion Criteria:

* people with skin problems in the head and neck area that that made the examination impossible
* previous head and neck surgeries and traffic injuries
* coagulation disorders or taking medications that reduce blood coagulability
* venous thrombosis in the neck area
* sensory disorders
* dislocation of the jaw in the past
* taking painkillers 12 hours before starting the study
* being under orthodontic or physiotherapeutic treatment focused on TMJ dysfunctions

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Students from Poland
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Pressure sensitivity | for each participant duration of test is about 30-40 minutes
  Algometer measurements on the upper fibers of the trapezius, levator scapula, sternocleidomastoid and rectus capitis posterior major

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for Rehabilitation, Poznan, Greater Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Sensitive data, maybe available on reasonable request